CLINICAL TRIAL: NCT00190151
Title: Pharmacokinetic/Pharmacodynamic Parameters Associated With the Emergence of Resistance to Ciprofloxacin in Human Commensal Flora
Brief Title: Parameters Associated With the Emergence of Resistance to Ciprofloxacin in Human Commensal Flora
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department Clinical Research of Developpement
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P031007
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2005-09

CONDITIONS: Healthy Volunteers
Keywords: ciprofloxacin; commensal flora; resistance; Pharmacokinetic
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ciprofloxacin

SUMMARY:
Bacterial resistance to antibiotics has been a growing therapeutic problem since the late 1980s. Resistant strains of pathogenic bacteria can arise through initial selection of resistant strains in the commensal flora. The emergence of fluoroquinolone resistance in the commensal flora will be assessed in 48 healthy volunteers receiving variable doses of ciprofloxacin during 14 days. Emergence of resistance will be correlated to pharmacokinetic characteristics of ciprofloxacin.

DETAILED DESCRIPTION:
Pharmacokinetic/Pharmacodynamic Parameters Associated With the Emergence of Resistance to Ciprofloxacin in Human Commensal Flora Bacterial resistance to antibiotics has been a growing therapeutic problem since the late 1980s. Resistant strains of pathogenic bacteria can arise through initial selection of resistant strains in the commensal flora. The emergence of fluoroquinolone resistance in the commensal flora will be assessed in 48 healthy volunteers receiving variable doses of ciprofloxacin during 14 days. Emergence of resistance will be correlated to pharmacokinetic characteristics of ciprofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-09; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of bacterial resistance in commensal flora

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic relationship

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fantin, Study Chair — Hôpital Beaujon, 100 boulevard du Général Leclerc, 92110 Clichy, France; Xavier Duval, Principal Investigator — Hôpital Bichat Claude Bernard, 48 rue Henri Huchard, 75877 Paris Cedex 18, France
Locations (1):
- Hôpital Bichat Claude Bernard, 46 rue Henri Huchard, Paris, France

REFERENCES:
- [Derived] de Lastours V, Maugy E, Mathy V, Chau F, Rossi B, Guerin F, Cattoir V, Fantin B; CIPHARES Study Group. Ecological impact of ciprofloxacin on commensal enterococci in healthy volunteers. J Antimicrob Chemother. 2017 Jun 1;72(6):1574-1580. doi: 10.1093/jac/dkx043. PMID 28333351
- [Derived] de Lastours V, Cambau E, Guillard T, Marcade G, Chau F, Fantin B. Diversity of individual dynamic patterns of emergence of resistance to quinolones in Escherichia coli from the fecal flora of healthy volunteers exposed to ciprofloxacin. J Infect Dis. 2012 Nov;206(9):1399-406. doi: 10.1093/infdis/jis511. Epub 2012 Aug 28. PMID 22930806
- [Derived] Fantin B, Duval X, Massias L, Alavoine L, Chau F, Retout S, Andremont A, Mentre F. Ciprofloxacin dosage and emergence of resistance in human commensal bacteria. J Infect Dis. 2009 Aug 1;200(3):390-8. doi: 10.1086/600122. PMID 19563257